CLINICAL TRIAL: NCT06883214
Title: Deciphering the Functional Role of a Three-miRNA Signature in Glioma: From Molecular Mechanisms to Potential Clinical Application
Brief Title: Three miRNA Signatures in Glioma: From Molecular Mechanisms to Potential Clinical Application
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of Roma La Sapienza (Other); San Camillo Hospital, Rome (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Neuromed IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: RS1821/23
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individual overexpression of the three miRNAs negatively affects cell viability and proliferation mainly in grade III IDH-wild type cells, while in higher grade cells, the effect is more pronounced when the entire signature is overexpressed, individual and combined overexpression of the signature members is able to determine a significant reduction in both migration and invasion. Therefore, ectopic expression of the miRNAs identified by us has a negative impact on cell viability, proliferation and apoptosis, but above all on migration and invasion.

DETAILED DESCRIPTION:
Decipher the impact and functional role of the signature formed by miR-1-3p, miR-26a-1-3p and miR-487b-3p on glioma biology. The functional role of the miRNAs of the signature will be assessed with gain/loss of function strategies, using primary glioma cells derived from patients with native IDH-wild type or mutated status. To set up the system we will start the study using glioma cell lines derived from patients already well characterized from a molecular and immunohistochemical point of view following the criteria reported by the new update of the 2016 WHO classification of tumors of the central nervous system. Furthermore, the involvement of the signature in the response to treatment will be evaluated. Despite the application of the most recent treatment protocols, the prognosis of patients with glioma remains unfavorable especially for patients with grade 4 glioma IDH-wild type in which resistance to radiotherapy and temozolamide contributes significantly to the negative outcome. Since it has been reported that some miRNAs can promote chemosensitization on a wide variety of tumors, including gliomas, the involvement of the miRNA signature in the response to treatment of these tumors will be studied. Cellular sensitivity to radiotherapy and temozolamide will be evaluated by dose-response curves in cell lines and primary cells derived from both IDH-wild type and IDH-mutated patients.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of glioma;
* no concomitant primary tumor;
* no metastatic disease;
* availability of surgical material/tissue;
* written informed consent.

Exclusion Criteria:

* histological diagnosis of non-glial tumor;
* patients with concomitant other solid tumors;
* metastatic disease;
* no surgical material/tissue available;
* HIV seropositivity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tissue samples from patients with glioma
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-01-17 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
Dose-response curves | 36 months
  Cellular sensitivity to radiotherapy and temozolamide will be assessed by dose-response curves in both IDH-wild type and IDH-mutated patient-derived cell lines and primary cells.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy